CLINICAL TRIAL: NCT01580501
Title: Functional Muscle Ischemia and PDE5 Inhibition in Duchenne Muscular Dystrophy: Acute Dosing Study
Brief Title: PDE Inhibitors in DMD Study (Acute Dosing Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ron Victor, Associate Director of the Hypertension Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 27521
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tadalafil and Sildenafil — PDE-5 Inhibitor; Low dosages will be 0.5mg/kg and high dosages will be 1.0mg/kg
  Other Names: Tadalafil/Cialis; Sildenafil/Viagra

SUMMARY:
PDE5A inhibition, which boosts NO-cGMP signaling, will relieve functional muscle ischemia and restore normal blood flow regulation (i.e., functional sympatholysis) during exercise in boys with DMD. The investigators specific aim is to perform an efficient dose-titration study to inform the design of a randomized multicenter trial of PDE5A inhibition for clinical skeletal muscle and cardiac endpoints.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is a rare, progressive and fatal muscle disease affecting boys and accounts for 80% of muscular dystrophy cases. Tadalafil and sildenafil are medications approved by the FDA for the treatment of erectile dysfunction and pulmonary hypertension. This class of medication improves muscle blood flow in a mouse model of muscular dystrophy, but their benefit to boys with DMD is unknown. The purpose of this study is to perform an efficient dos-titration study to inform the design of a randomized multicenter trial of PDE5A inhibition for clinical skeletal muscles and cardiac endpoints.

The investigators will enroll boys with DMD between the ages of 7 and 15 years who are ambulatory and without clinical heart failure. Participants will undergo five visits and one follow up phone call over a one month period. The initial visit will include a medical history, physical exam, echocardiogram, and blood draw to determine eligibility for the study.

Eligible boys will be given two different study drugs: sildenafil and tadalafil. At the first set of visits, the boys will take a low dose (0.5mg/kg) of the sildenafil for the first day and a high dose (1.0mg/kg) for the second day. Blood will be drawn at specific timepoints to obtain drug levels (15 minutes, 30 minutes, 1-, 2-, 4-, and 8-hours post dosing). The boys will be asked to return approximately one week later for the second set of visits to take the other study drug, tadalafil. The boys will be take a low dose (0.5mg/kg) of tadalafil for the first day and a high dose (1.0mg/kg) for the second day. Again, blood will be drawn at specific timepoints.

All eligible subjects will be given both open-label sildenafil initially and then tadalafil.

There will be five clinic visits (screening visit, two sets of medication visits) and one follow up phone call. For these visits, boys will undergo an arm blood flow and hand grip exercise protocol. In this procedure, blood flow and oxygen delivery to the forearm muscles will be measured (noninvasively) before and during application of lower body negative pressure at rest and during handgrip exercise. Lower body negative pressure stimulates the blood flow changes that normally occur when a person sits up after lying down. During the medication visits, boys will have a saline lock inserted in a vein in their arm to obtain blood for study drug levels.

A one week follow-up telephone call will be done to check for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of DMD confirmed by muscle biopsy or DNA analysis
2. age 7-15y
3. ambulatory
4. no clinical evidence of heart failure

Exclusion Criteria:

1. hypertension, diabetes, or heart failure by standard clinical criteria
2. elevated BNP level (>100 pg/ml)
3. LVEF < 50%
4. non-ambulatory
5. cardiac rhythm disorder, specifically: rhythm other than sinus, SVT, atrial fibrillation, ventricular tachycardia
6. continuous ventilatory support
7. liver disease
8. renal impairment
9. contraindications to sildenafil (use of nitrates, alpha-blockers, CYP3A inhibitors, amlodipine, or other PDE5A inhibitors)

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pre vs. post treatment change in functional sympatholysis by NIR for each dose of each drug.
  Measured by the decrease in muscle tissue oxygenation (near infrared spectroscopy) and blood flow (Doppler ultrasound) evoked by reflex sympathetic activation in exercising forearm muscle.

SECONDARY OUTCOMES:
Sympatholysis measured by brachial artery Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States